CLINICAL TRIAL: NCT06528288
Title: Opioid Usage and Patient Reported Outcome Comparison Following Erector Spinae Plane Block or Subcutaneous Anesthetic in Spinal Fusion Procedures
Brief Title: Effects of Erector Spinae Plane Block on Postoperative Pain Following Lumbar Fusion Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Michael Stauff, Assistant Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00001297
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Fusion of Spine, Lumbar Region; Anesthesia, Local; Pain, Postoperative; Opioid Use
Keywords: Erector Spinae Plane Block; Spinal Fusion; Patient Reported Outcomes; Opioid Usage
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be masked to the treatment arm. The research team (outcomes assessors) involved in evaluation of subjects will be blinded to the treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erector Spinae Plane Block (Experimental): An erector spinae plane block (ESPB) will be administered prior to the surgical procedure, but after the patient receives general anesthesia. The injection will consist of 10 mL of saline, 20 mL of liposomal bupivacaine, and 30 mL of bupivacaine. This will be injected along the erector spinae fascial plane at the surgical levels. Fluoroscopy will be used for guidance during the injection.
  Interventions: Procedure: Erector Spinae Plane Block
- Subcutaneous Anesthesia (Active Comparator): A subcutaneous anesthesia injection will be administered after the surgery has been completed, but while the patient is under general anesthesia. The injection will consist of 10 mL of saline, 20 mL of liposomal bupivacaine, and 30 mL of bupivacaine. This will be injected around the surgical incision, subcutaneously.
  Interventions: Procedure: Subcutaneous Anesthesia

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — The erector spinae plane block (ESPB) is a method for injecting local anesthesia to reduce pain related to a surgical procedure. The anesthesia is theorized to spread along the paraspinal fascia and anesthetize a larger area, resulting in patients reporting less pain and using less opioids postoperatively.
  Arms: Erector Spinae Plane Block
Procedure: Subcutaneous Anesthesia — Subcutaneous anesthesia injection involves placement of local anesthesia under the skin around the surgical incision. This is thought to reduce pain from the incision site postoperatively.
  Arms: Subcutaneous Anesthesia

SUMMARY:
The purpose of this study is to determine if the method for injecting local anesthesia affects patients' pain and opioid usage after surgery. The investigators will compare subcutaneous anesthesia, injections of anesthesia under the skin, to a method called erector spinae plane block (ESPB). An ESPB injection involves placing local anesthesia along the muscles and bones in the back, using a special type of x-ray called fluoroscopy for guidance. The Investigators will use patient reported outcomes (PROs) and track subjects' opioid usage to find out if there is a difference between ESPB and subcutaneous anesthesia. The investigators hypothesize that patients who get ESPB injections will use less opioids and report less pain after lumbar fusion surgery compared to patients who receive subcutaneous anesthesia injections.

ELIGIBILITY:
Inclusion Criteria:

* The individual has signed and dated a study specific informed consent form approved by the Institutional Review Board at UMMHC.
* The individual is at least 18 years of age.
* The individual is skeletally mature (over the age of 18).
* The patient is scheduled for a one or two level lumbar spinal fusion.

Exclusion Criteria:

* Patients unable to consent for themselves.
* Pregnant women.
* Non-English speaking subjects.
* Prisoners.
* Spinal fusion procedures for a diagnosis of fracture, tumor, and/or infection.
* Patients who have used greater than 150 morphine milligram equivalents of opioids in the month prior to their operation.
* Patients with a body mass index (BMI) of 40 or greater.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
MOS 36 Item Short Form Health Status Survey (SF-36) | 3 months
  Questionnaire related to a patient's general health, bodily pain, physical function, and mental health. Scoring includes eight scaled scores, which are the weighted sums of the questions in their section. Scales are converted into a 0-100 scale. The lower the score the more disability. The higher the score the more functionality and therefore indicating better outcome.
Oswestry Disability Index | 3 months
  Questionnaire related to a patient's back pain and its impact on their day-to-day activities. There are 10 questions, each weighted from 0-5 points. The point total of each question is added together to give a final scaled score ranging from 0-50. Lower scores near 0 are indicative of better outcome and less disability, while higher scores near 50 indicate worse outcomes and more disability.
Postoperative Opioid Usage | 2 weeks
  This is a tracking sheet for the amount of opioid medications used in the first 2 weeks of postoperative recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stauff, MD, Principal Investigator — UMass Chan Medical School
Locations (1):
- UMass Chan Medical School/UMass Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be shared after deidentification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available immediately following publication and will remain available for six (6) years.
Access Criteria: The data will be provided to researchers who provide a methodologically sound proposal.